CLINICAL TRIAL: NCT06390410
Title: A Pharmacokinetic Study of Simufilam in Subjects With Impaired Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cassava Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PTI-125-11
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Hepatic Insufficiency
MeSH Terms: conditions — Hepatic Insufficiency | interventions — Simufilam

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Moderate Hepatic Impairment (Experimental)
  Interventions: Drug: Simufilam
- Healthy Volunteer (Experimental)
  Interventions: Drug: Simufilam
- Mild Hepatic Impairment (Experimental)
  Interventions: Drug: Simufilam

INTERVENTIONS:
Drug: Simufilam — 100 mg PTI-125

SUMMARY:
Evaluate simufilam levels in the blood of hepatically impaired individuals compared to Healthy individuals of similar demographics

DETAILED DESCRIPTION:
This is a Phase I, open label, single-dose study of simufilam 100 mg. Up to 34 subjects may be enrolled; 10 subjects with moderate hepatic impairment, 10 healthy volunteers with normal hepatic function (with the potential of 4 more), and if needed 10 subjects with mild hepatic impairment. Both males and females will be enrolled. The study will be conducted in 2 groups (with the potential of a third) assigned based on degree of hepatic impairment as follows:

up to 10 subjects with moderate hepatic impairment (Child-Pugh score of 7-9) up to 10 health volunteers (matched to each hepatic impairment severity group)

If needed up to 10 subjects with mild hepatic impairment (Child-Pugh score of 5-6), and an additional 4 healthy volunteers if needed to match the mild group

ELIGIBILITY:
Inclusion Criteria:

* The subject is willing and able to speak, read, and understand English and is willing to provide written informed consent.
* Male or female subjects between 18 and 75 years of age, inclusive.
* The subject has a body mass index (BMI) within 18-40 kg/m2.
* The subject must have renal function that is normal or consistent with mild renal insufficiency.
* The subject has normal/acceptable mental status for study participation in the opinion of the Investigator.
* Male subjects and female subjects of childbearing potential must agree to their respective birth control requirements. Females of non-childbearing potential must satisfy the definition of permanent sterility or postmenopausal status
* The subject must agree to comply with the drawing of blood samples for the pharmacokinetics (PK) assessments.
* The subject is willing and able to comply with all testing and requirements defined in the protocol.
* The subject is willing and able to remain at the study site unit for the duration of the study.
* The subject must be negative for the COVID virus at both the Screening Visit and the Check-In Visit.

Additional inclusion criteria specific for subjects with normal hepatic function:

* The subject with normal hepatic function is in reasonably good health, determined by no clinically significant findings from medical history, physical examination, 12-lead electrocardiogram (ECG), vital sign measurements, and clinical laboratory evaluations in the opinion of the Investigator and/or Medical Monitor.

Additional inclusion criteria specific for subjects with hepatic impairment:

* Subjects with hepatic impairment with other stable, chronic medical conditions (e.g., hypertension, hyperlipidemia, diabetes) may be included if, in the opinion of the Investigator and Medical Monitor, the abnormality will not significantly alter the disposition of the drug and will not interfere with interpretation of the data.
* The subject with moderate or mild hepatic impairment has been diagnosed at least 6 months prior to Screening.

  * Moderate: Child-Pugh Class B (7 to 9 points)
  * Mild: Child-Pugh Class A (5 to 6 points) (if a decision is taken to enroll)
* The subject with hepatic impairment has clinical laboratory tests that are considered clinically stable and consistent with the subject's disease, in the opinion of the investigator.

Exclusion Criteria:

* The subject has a clinically significant electrocardiogram (ECG) abnormality including, but not necessarily limited to, a confirmed QT interval by the Fridericia correction formula (QTcF) > 470 msec (females) or > 450 msec (males) based on WHO 2016 guidelines.
* The subject has had a clinically significant illness within 30 days prior to the Screening Visit.
* The subject has a medically significant comorbid illness that would impact the successful conduct of the study or achieving its objectives in the opinion of the Investigator and/or Medical Monitor.
* The subject has used a known strong CYP2C19 inhibitor (fluconazole, fluoxetine, fluvoxamine or ticlopidine) or inducer (rifampin) within 28 days prior to admission, or 5 half-lives (whichever is longer).
* The subject has consumed alcohol, grapefruit, grapefruit juice, caffeine- or xanthine-containing products within 72 hours before dosing or intends to use any of these products during the study.
* The subject has smoked more than 10 cigarettes per day on average for the past 6 months.
* The subject has a history of substance abuse within 12 months of the Screening Visit.
* The subject tests positive on the urine drug screen for drugs of abuse at either the Screening Visit or the Check-In Visit (Note - Subjects with hepatic impairment who are prescribed medications assessed in the urine drug screen [e.g, opiates, benzodiazepines] need not be excluded based on a positive urine drug screen).
* The subject has a positive ethanol breath test at either the Screening Visit or the Check-In Visit.
* The subject has a history of regular alcohol consumption defined as greater than 7 drinks per week for women and 14 drinks per week for men within six months prior to the Screening Visit.
* The subject has a positive serum hepatitis B surface antigen test at the Screening Visit.
* The subject has a positive human immunodeficiency virus (HIV) test at the Screening Visit.
* The subject is pregnant or breastfeeding.
* The subject has received an investigational drug within 30 days or five half-lives - whichever is longer - prior to Study Day 1.
* The subject has previously received simufilam.
* The subject has donated or lost a significant volume of blood (>500 mL) within a 90 day period prior to the Screening Visit. This does not include plasma donation.
* Subjects with poor peripheral venous access.
* Subjects who, in the opinion of the Investigator (or designee), should not participate in this study.

Additional exclusion criteria specific for subjects with normal hepatic function:

* The subject with normal hepatic function has or has had hepatitis C, as confirmed by a positive hepatitis C virus (HCV) antibody test at the Screening Visit.
* The subject with normal hepatic function has used prescription or over the counter (OTC) medication within 7 days prior to the Check-In visit, or intends to use any prescription or OTC medication during the study, with the following exceptions:

  * Hormonal contraceptives,
  * Over-the-counter analgesics, stool softeners, and/or multivitamins up to 48 hours prior to study drug administration.

Additional exclusion criteria specific for subjects with hepatic impairment:

* The subject with hepatic impairment has used prescription or OTC medication within 7 days prior to the Check-In Visit except for the management of their hepatic impairment or stable, chronic medical conditions. Such medications must have a stable dose regiment and be approved by the Medical Monitor (Note - over-the-counter analgesics, stool softeners, and/or multivitamins up to 48 hours prior to study drug administration are acceptable).
* The subject with hepatic impairment has a hemoglobin level < 9.0 (g/dL) or a platelet count < 35×109/L.
* The hepatically impaired subject with type 2 diabetes on standard oral medication has a HbA1C > 9.5% at either the Screening Visit or the Check-In Visit (Note - use of insulin is not acceptable).
* The subject with hepatic impairment who has a positive hepatitis C virus (HCV) antibody test also has a positive HCV RNA test (that confirms chronic infection upon reflex testing).
* The subject with hepatic impairment has evidence of active hepatic encephalopathy > Grade 2 or history of >Grade 2 within the last 6 months. Subject with a history of > Grade 2 hepatic encephalopathy more than 6 months prior to Screening and who currently receives medication for treatment may be allowed, but should be assigned the pre-treatment Child-Pugh score of hepatic encephalopathy.
* The subject with hepatic impairment has acute hepatitis, severe ascites (defined by the need for frequent paracentesis), hepatocellular carcinoma, current unstable hematological condition, recent upper gastrointestinal bleed, surgical portosystemic shunts, or evidence of hepatorenal syndrome.
* The subject with hepatic impairment has history of pancreatitis within 4 months of Screening.
* The subject with hepatic impairment has had a liver transplant prior to Screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2024-06-26 (Actual); Primary Completion 2024-12-07 (Actual); Study Completion 2024-12-07 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve; moderate vs. normal and mild vs. normal | 5 Days
  Area Under the Curve of simufilam concentration in plasma in Moderate and Mild Impairment vs. Normal (each separately)
Concentration max; moderate vs. normal and mild vs. normal | 5 Days
  Maximum simufilam concentration in plasma in Moderate and Mild Impairment vs. Normal (each separately)
Time max; moderate vs. normal and mild vs. normal | 5 Days
  Time to maximum simufilam concentration in plasma in Moderate and Mild Impairment vs. Normal (each separately)
Half-life; moderate vs. normal and mild vs. normal | 5 Days
  Half-life of simufilam concentration in plasma in Moderate and Mild Impairment vs. Normal (each separately)
Elimination rate constant; moderate vs. normal and mild vs. normal | 5 Days
  Elimination rate constant of simufilam concentration in plasma in Moderate and Mild Impairment vs. Normal (each separately)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Orange County Research Center, Lake Forest, California
  - Clinical Pharmacology of Miami, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida